CLINICAL TRIAL: NCT00562081
Title: Evaluation of an Internet-based Approach to Long-term Treatment of Asthma.
Brief Title: The Virtual Asthma Clinic
Acronym: VAC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment.
Sponsor: University of Alberta (Other)
Collaborators: ASTHMA C Project (Unknown); AstraZeneca (Industry); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M-2394
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2009-01

CONDITIONS: Asthma
Keywords: asthma; Virtual Asthma Clinic; metabolites; asthma education
MeSH Terms: conditions — Asthma | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Patient does not have 24/7 access to a Certified Asthma Educator.
  Interventions: Behavioral: Education
- 2 (Active Comparator): Patient has 24/7 access to a Certified Asthma Educator.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — 24/7 access to a Certified Asthma Educator
  Arms: 2
Behavioral: Education — Patient does not have 24/7 access to a Certified Asthma Educator.
  Arms: 1

SUMMARY:
Patients with asthma can be effectively treated using an Internet-based management system as demonstrated by:

1. Physician utilization (emergency department visits and unscheduled physician visits).
2. Health-related quality of life scores.
3. Global health care costs.
4. Frequency of severe exacerbations and time to first exacerbation.
5. Asthma control days.
6. Patient education.

Effective patient education will be associated with decreased markers of inflammation and improved indices of airways function.

DETAILED DESCRIPTION:
Over a one-year period, we will evaluate specific outcomes related to the use of the internet-based asthma treatment plans. Patients identified by their physician as candidates for the study will be screened by the CAE. All subjects will be provided with an information sheet and will be asked to sign an informed consent. All subjects asthma treatment will be reviewed for adequacy of medical management (as defined by the Canadian Consensus Guidelines for Asthma Care) and may have treatment adjusted by one of the study physician specialists to ensure compliance with guideline-based best practice if necessary

Following obtaining consent, all subjects will receive identical standardized education. This will include: review of medications and inhaler device technique, review any environmental triggers, and generate a written action plan. All subjects will receive a peak flow meter and will be instructed in its use. All subjects will undergo baseline pulmonary function tests if they have not had one conducted in the previous six months that will include flow-volume loops pre and post bronchodilator. Subjects that do not demonstrate a 12% improvement in FEV1 post bronchodilator will also have a methacholine challenge test to assess airway hyperreactivity. A urine sample will be obtained and frozen for subsequent NMR spectroscopy. Standard demographic information will be obtained from all subjects including smoking status, age, education status, and weight assessed as BMI. Subjects successfully completing screening tests and fulfilling inclusion and exclusion criteria will be randomly allocated to either to the active therapy using the Internet site, or to a placebo therapy using a web-based intervention. Randomization will occur using an internet based program created by the EPICORE Centre at the University of Alberta.

All subjects will be given an individualized access code and the website address and will receive a brief demonstration of the website. Following initial log-on to the website the subject's in the intervention group will have their asthma profile reviewed daily by a Certified Asthma Educator (CAE). Patients who do not log-on to the website within 1 week of randomization will be contacted by telephone. The intervention group will have access to the full version of the website with access to the CAE and they will be expected to enter daily symptoms, evening and morning peak flows and medication use under their subject profile. Patients who consent but do not log-on despite additional telephone contact will be deemed as an immediate compliance failure. Otherwise patients' individual profiles will be evaluated until the end of the 12-month period. Non-compliance to the asthma management program will be defined as:

1. Failure to enter any information for 7 consecutive days for patients experiencing poor asthma control in the preceding 2 weeks.
2. Failure to enter any information for 14 consecutive days for patents experiencing good asthma control in the preceding 2 weeks. This point will be deemed the time to compliance failure.

The internet-based system will utilize a secure website to deliver the following to the intervention group: 1) ongoing patient education, 2) regular feedback regarding significance of symptoms, 3) regular feedback regarding significance of peak flows, and 4) a written action plan. Patients will also have their individual files monitored regularly by a CAE. Finally patients in the intervention group will have on-line access to an asthma educator through a secure email system.

The placebo web-based intervention will include basic patient information on asthma and asthma management; however will not include an interactive component. They would not have personalized information tracked on the asthma management website, however they will be asked to complete the outcome measurements at regularly scheduled intervals online. All subjects will be sent regular email reminders to continue to log into the program and complete the outcome measures. These reminders will be sent at regular intervals and include basic information on asthma to encourage participation.

All patients will be requested to provide their Alberta Health Care Insurance Plan Number to allow access to their individualized health care utilization data from Capital Health and the Calgary Regional Health Authority. In particular, clinic visits; emergency room visits; and hospitalization data will be requested from the health regions. Patients will also be asked to provide a copy of their prescription records for the duration of the study. All data will be entered into a SPSS database and will be analyzed using this and other statistical programs. Data analysis will be conducted by EPICORE at the University of Alberta.

All subjects will be monitored via website for one year. All subjects will be asked to complete the 15D and AQLQ at baseline, six months post enrollment and 12 months post enrollment. Additionally, they will be asked to complete the Weekly Survey every two months. The intervention group only will be asked to complete the symptom survey at each login, as it is used primarily for clinical reasons by the CAE. All subjects will have seven days to complete and submit the outcome measures and reminders will be sent via email every second day. If a subject fails to complete the measurements within the seven-day period, they will receive a phone call reminder. Subjects will be asked to return 12 months post enrollment to the clinic for repeated spirometry testing and a second urine sample collection. No additional office visits are anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of asthma at the time of enrolment.
2. The forced expiratory volume in one second (FEV1) at base line will be at least 50 percent of the predicted value.
3. Evidence of at least 12% increase in FEV1 following inhaled bronchodilator or airway hyperreactivity as defined by a standard methacholine challenge study.

Exclusion Criteria:

1. Concurrent disease likely to require regular physician contact (e.g. congestive heart failure).
2. A separate diagnosis or other pulmonary disease (e.g. pulmonary fibrosis or chronic bronchitis).
3. An inability to access the Internet on a regular basis.
4. Inability or unwillingness to give informed consent or to complete online health related quality of life questionnaires.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Emergency department visits and unscheduled physician visits | One year.
Good asthma control days | One year.
Time to first severe exacerbation | One year.

SECONDARY OUTCOMES:
Morning peak expiratory flow | One year.
Percentage of days with symptoms | One year.
Percentage of nights with asthma awakenings | One year.
Number of rescue inhalations per week | One year.
Health related quality of life scores | One year.
Markers of inflammation: Airway hyperreactivity, Urine metabolic activity | One year.
Health economic assessment: Frequency of direct health care provider contacts, Medications, Travel costs associated with medical care, Over the counter medications e. Internet/computer costs | One year.

CONTACTS AND LOCATIONS:
Overall Officials: Irvin Mayers, MD, FRCPC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada